CLINICAL TRIAL: NCT05526755
Title: An Open-label, Single-arm, Phase II, Multinational, Multicentre Study to Assess the Efficacy and Safety of 5 Years of Osimertinib in Participants With EGFRm-positive Stage II-IIIB NSCLC, Following Complete Tumour Resection With or Without Adjuvant Chemotherapy
Brief Title: A Study of 5 Years of Adjuvant Osimertinib in Completely Resected Epidermal Growth Factor Receptor Mutation (EGFRm) Non-small Cell Lung Carcinoma (NSCLC)
Acronym: TARGET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5162C00048; 2023-508740-21-00 (Registry Identifier: CTIS (EU)); 2021-003024-33 (EudraCT Number)
Record Dates: First submitted 2022-09-01; First posted 2022-09-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Stage II-IIIB Non-small Cell Lung Carcinoma
Keywords: Stage II-IIIB Non-small Cell Lung Cancer; Adjuvant osimertinib; Adjuvant chemotherapy
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental): Participants will receive osimertinib (AZD9291).
  Interventions: Drug: Osimertinib 80 mg/40 mg

INTERVENTIONS:
Drug: Osimertinib 80 mg/40 mg — Participants will receive osimertinib (80 mg or 40 mg orally, once daily).
  Other Names: AZD9291; TAGRISSO™

SUMMARY:
To assess the efficacy and safety of osimertinib in participants with EGFRm positive stage II-IIIB NSCLC, following complete tumour resection with or without adjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a phase 2 open-label study to assess the efficacy and safety of osimertinib in participants with stage II-IIIB NSCLC with sensitising EGFR mutations. The study is designed to evaluate 5 years of adjuvant osimertinib therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged at least 18 years.
2. Histologically confirmed diagnosis of primary NSCLC on predominantly non-squamous histology.
3. Magnetic Resonance Imaging (MRI) or contrast computed tomography (CT) scan of the brain.
4. Participants must be classified post-operatively as Stage II, IIIA, or IIIB on the basis of surgical pathologic criteria.
5. Confirmation by the local laboratory that the tumour harbours one of the two common EGFR mutations (Ex19del, L858R), either alone or in combination with other EGFR mutations including de novo EGFR mutation resulting in substitution of threonine with methionine at amino acid position 790 in exon 20 of EGFR (T790M) or uncommon EGFR mutations G719X, S768I, and L861Q, either alone, in combination with each other, or in combination with other uncommon EGFR mutations (excluding all exon 20 insertions) (Uncommon EGFRm Cohort).
6. Complete surgical resection of the primary NSCLC is mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumour.
7. Complete recovery from surgery and standard post-operative therapy (if applicable) at start of study intervention.
8. World Health Organisation Performance Status of 0 to 1.
9. Female participants must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of childbearing potential.
10. Male participants must use effective barrier contraception.

Exclusion Criteria:

1. Major surgery (including primary tumour surgery, excluding placement of vascular access) within 4 weeks prior to the first dose of study drug.
2. Participants currently receiving medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 weeks prior to first dose).
3. Participants who have had only segmentectomies or wedge resections.
4. History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer, or other solid tumours curatively treated with no evidence of disease for > 5 years before the start of study intervention.
5. Treatment with any of the following:

   * Pre-operative or post-operative or planned radiation therapy for the current lung cancer.
   * Pre-operative (neo-adjuvant) platinum-based or other chemotherapy.
   * Any prior anti-cancer or immunological therapy, including investigational therapy, for treatment of NSCLC other than standard platinum-based doublet post-operative adjuvant chemotherapy.
   * Prior treatment with neoadjuvant or adjuvant EGFR tyrosine kinase inhibitor (TKI).
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
7. Any of the following cardiac criteria:

   * Mean resting corrected QT (QTc) interval > 470 msec, obtained from 3 electrocardiograms (ECGs).
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events.
   * Heart failure, congenital long QT interval (QT) syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes (TdP).
8. Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.
9. Inadequate bone marrow reserve or organ function.
10. Women who are breastfeeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2029-11-22 (Estimated); Study Completion 2029-11-22 (Estimated)

PRIMARY OUTCOMES:
Estimate the Efficacy of Osimertinib as Measured by Disease Free Survival (DFS) [Common EGFRm Cohort]. | From date of first dose until date of disease recurrence or death (by any cause in the absence of recurrence), up to approximately 5 years. Assessed at 5 years.
  Defined as time from date of first dose until disease recurrence, or death due to any cause in the absence of recurrence.

SECONDARY OUTCOMES:
Disease Free Survival Rate at 3, 4 and 5 Years (Uncommon EGFRm Cohort) | From date of first dose until date of disease recurrence or death (by any cause in the absence of recurrence), up to approximately 5 years. Assessed at 3 years, 4 years, and 5 years.
  Defined as the proportion of participants alive and disease free at 3, 4, and 5 years.
DFS Rate at 3 and 4 Years (Common EGFRm Cohort) | From date of first dose until date of disease recurrence or death (by any cause in the absence of recurrence), up to approximately 5 years. Assessed at 3 years, and 4 years.
  Defined as the proportion of participants alive and disease free at 3, and 4 years.
Overall Survival (OS) [Common EGFRm Cohort] | From date of first dose until the date of death due to any cause, up to approximately 5 years. Assessed at 3 years, 4 years, and 5 years.
  Defined as time from date of first dose until the date of death due to any cause.
Safety and tolerability in overall population (Common EGFRm Cohort and Uncommon EGFRm Cohort) | From date of first dose up to approximately 5 years
  Adverse Events (AEs) graded by CTCAE version 5.0.
Recurrence events in overall population (Common EGFRm Cohort and Uncommon EGFRm Cohort) | From date of first dose up to approximately 5 years
  Local/regional, or distant recurrence events assessed.

CONTACTS AND LOCATIONS:
Locations (46):
- United States (3):
  - Research Site, Santa Rosa, California
  - Research Site, Las Vegas, Nevada
  - Research Site, White Plains, New York
- Research Site, Hong Kong, Hong Kong
- Italy (11):
  - Research Site, Avellino
  - Research Site, Brescia
  - Research Site, Lecce
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Peschiera del Garda
  - Research Site, Reggio Emilia
  - Research Site, Sondrio
  - Research Site, Terni
  - Research Site, Udine
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Kuching
- Philippines (3):
  - Research Site, Cebu
  - Research Site, Manila
  - Research Site, Quezon City
- Research Site, Singapore, Singapore
- South Korea (8):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Granada
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Songkhla
- United Kingdom (2):
  - Research Site, London
  - Research Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual participant-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Soo RA, de Marinis F, Han JY, Ho JC, Martin E, Servidio L, Sandelin M, Popat S. TARGET: A Phase II, Open-Label, Single-Arm Study of 5-Year Adjuvant Osimertinib in Completely Resected EGFR-Mutated Stage II to IIIB NSCLC Post Complete Surgical Resection. Clin Lung Cancer. 2024 Jan;25(1):80-84. doi: 10.1016/j.cllc.2023.09.005. Epub 2023 Oct 4. PMID 37914594